CLINICAL TRIAL: NCT05125354
Title: A Retrospective Analysis to Evaluate Long Term Outcomes of Squamous Cell Carcinoma Patients Previously Treated With Alpha Diffusing Alpha-emitters Radiation Therapy
Brief Title: A Retrospective Analysis to Evaluate Long Term Outcomes of SCC Patients Previously Treated With Alpha DaRT
Status: Completed | Type: Observational
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP-SCC-02
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-10

CONDITIONS: Squamous Cell Carcinoma; DaRT Treated Patients
Keywords: Squamous Cell Carcinoma; Alpha Radiation
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of long-term efficacy outcomes of patients previously treated with the Alpha DaRT seeds for management of their malignancy following initial response.

DETAILED DESCRIPTION:
Medical records of patients that previously underwent the Alpha DaRT treatment will be reviewed by an authorized staff member.

Evaluation of long-term outcomes of patients previously treated with the Alpha DaRT seeds for management of their malignancy following initial response. These outcomes include:

* Safety - assessment of late onset of Alpha DaRT related AE in patients treated with the Alpha DaRT seeds
* Efficacy -

  * assessment of local recurrence rates in patients who achieved initial complete response (CR) following the Alpha DaRT treatment
  * assessment of duration of response in patients who achieved initial CR following the Alpha DaRT treatment
  * assessment of survival status in patients treated with the Alpha DaRT seeds

ELIGIBILITY:
Inclusion Criteria:

* Patients previously treated with the Alpha DaRT seeds for management of either skin or oral cavity SCC
* Available information in medical charts and records (electronic or paper)

Exclusion Criteria:

None.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The medical records of patients previously treated with Alpha DaRT as part of the completed clinical trial "CTP-SCC-00" will be accessed to follow up with their status, if available.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 60 months following DaRT insertion
  Time from DaRT insertion to disease progression (according to RECIST V1.1) or death, whichever occurs first
Adverse Events (AE) | Up to 60 months following DaRT insertion
  Assessment of late onset of Alpha DaRT related AE

SECONDARY OUTCOMES:
Duration of Response | Up to 60 months following DaRT insertion
  Time from partial or complete response to the first disease progression according to RECIST V1.1
Overall Survival (OS) | Up to 60 months following DaRT insertion
  Time from DaRT insertion to death

CONTACTS AND LOCATIONS:
Overall Officials: Noga Kurman, MD, Principal Investigator — Davidof Cancer Institution at Rabin Medical Center Israel
Locations (2):
- Davidof Cancer Institution at the Rabin Medical Center Israel, Petah Tikva, Israel
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, Italy